CLINICAL TRIAL: NCT05871528
Title: HEROES Registry: Registry of Patients With Remote Posterior cErebral Hemorrhage Following Reperfusion Treatment in Ischemic Stroke in Catalonia
Brief Title: Registry of Patients With Remote Posterior cErebral Hemorrhage Following Reperfusion Treatment in Ischemic Stroke
Acronym: HEROES-CAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Germans Trias i Pujol Hospital (Other); Hospital del Mar (Other); Hospital de Granollers (Other); Hospital Arnau de Vilanova (Other); Parc Taulí Hospital Universitari (Other); Consorci Sanitari del Garraf (Other); Hospital de Sant Joan Despí Moisès Broggi (Other); Hospital Clinic of Barcelona (Other); University Hospital of Girona Dr. Josep Trueta (Network); Hospital Universitari de Bellvitge (Other); Hospital Vall d'Hebron (Other); Agència de Qualitat i Avaluació Sanitàries (Other Government)
Responsible Party: Sponsor
Other Study IDs: IIBSP-HER-2020-79
Record Dates: First submitted 2023-05-04; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Ischemic Stroke; Intracranial Hemorrhages; Hemorrhagic Transformation Stroke
Keywords: Ischemic stroke; Thrombolysis; Hemorrhagic transformation stroke; Secondary prevention
MeSH Terms: conditions — Ischemic Stroke; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No hemorrhagic transformation: Patients with ischemic stroke treated with intravenous thrombolysis and no hemorrhagic transformation (IH1 or IH2 are allowed)
- Local hemorragic transformation: Patients with ischemic stroke treated with intravenous thrombolysis and hemorrhagic transformation PH1 or PH2
- Remote hemorrhage: Patients with ischemic stroke treated with intravenous thrombolysis and remote hemorrhage in areas without evident ischemia (rPH)

SUMMARY:
Introduction Remote cerebral hemorrhage following reperfusion treatment in ischemic stroke is rare (1.3-3.7% of all treated strokes) and is associated with worse functional and vital prognosis. Multicenter observational studies suggest that amyloid angiopathy may be one of the main risk factors for remote hemorrhage. Currently, it is unknown what happens to those patients with remote hemorrhage beyond 3 months of follow-up in terms of risk/benefit balance when receiving antiplatelet or anticoagulant therapy, as well as from a cognitive point of view. Considering an analogy with amyloid angiopathy, the hypothesis is that those patients with remote hemorrhage have a higher risk of intracranial hemorrhage during follow-up when receiving stroke secondary prevention, and will also present greater cognitive deterioration during long-term follow-up.

Main Objectives

* To explore the frequency and risk factors for intracranial hemorrhage during follow-up of patients with remote cerebral hemorrhage.
* To explore the frequency and progression of cognitive deterioration during follow-up in patients with remote cerebral hemorrhage.

Methodology Observational, prospective, multicenter registry with a population-based case-control design of consecutive patients with remote hemorrhage following reperfusion therapy in acute ischemic stroke. Inclusion criteria: Diagnosis of ischemic stroke with age greater than or equal to 18 years who has remote cerebral hemorrhage after receiving reperfusion therapy in the acute phase. Exclusion criteria: Lack of basic data (age, sex, neuroimaging data) or telephone for follow-up. The cases will be those patients with remote hemorrhage. For each case included, 4 consecutive controls will be included (2 with local parenchymal hemorrhagic transformation and 2 without hemorrhagic transformation). The data will be filled out within the (Codi Ictus de CATalunya) CICAT registry form (currently mandatory in all stroke centers in Catalonia) to which additional variables will be added. Telephone follow-up will be conducted at 3, 12, and 24 months.

Main study variable:

* Any type of spontaneous or traumatic intracranial hemorrhage during a 24-month follow-up.
* Score on the "Short Informant Questionnaire" scale (a validated 17-question questionnaire to be conducted over the phone, where a score higher than 57 points indicates cognitive impairment).

Expected sample size during a 2-year recruitment period: 105-300 patients (considering the participating centers to date).

Additional information. This study is endorsed by the "Pla Director de la Malaltia Vascular Cerebral" in Catalonia.

Participating Centers. Participation offers have been sent to the 28 hospitals in the hospital network of Catalonia with the capacity to administer intravenous fibrinolysis. Positive responses have been received from 13 of them so far. In case the project is accepted by the (Comité Ético de Investigación Clínica) CEIC Sant Pau, the centers that have not responded will be contacted again to obtain their participation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the criteria for being a case (remote hemorrhage) or control according to the definition of Heidelberg hemorrhagic transformations
2. Age 18 or older
3. Definite diagnosis of ischemic stroke (intracranial large vessel occlusion, compatible lesion on neuroimaging)
4. Administration of a fibrinolytic drug associated or not with endovascular therapy (intravenous or local)
5. Availability of a control brain imaging before the first 36 hours from reperfusion treatment.

Exclusion Criteria:

* Lack of basic data (age, sex, follow-up neuroimaging, contact phone number for follow-up).

Ages: 18 Years to 102 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study outlines a four-step process to identify and select cases for a study on remote hemorrhages with or without local hemorrhagic transformation. The first step is to identify cases by evaluating control neuroimaging, and if there are doubts, investigators can seek consensus decision-making. The second step is to select four controls for each case, two without hemorrhagic transformation and two with type 2 hemorrhagic transformation. The third step involves completing the CICAT registry form and additional variables, some of which are optional. The fourth and final step is to conduct telephone follow-up at 3, 12, and 24 months to collect variables of interest in relation to the study's objectives.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Explore the frequency and risk factors of intracranial hemorrhage during follow-up in patients with remote cerebral hemorrhage | 24 months
  Describe the frequency, rate and adjusted hazard ratio

SECONDARY OUTCOMES:
Explore the frequency of ischemic stroke, intracerebral hemorrhage, intracranial hemorrhage, and any cerebrovascular event in patients with remote cerebral hemorrhage. | 24 months
  Describe the frequency, rate and adjusted hazard ratio
Investigate the net benefit of preventive treatment in patients with remote cerebral hemorrhage (composite of ischemic stroke and intracranial hemorrhage). | 24 months
  Evaluate the rate and adjusted hazard ratio of ischemic and hemorrhagic events
Explore the socio-functional status of patients with remote cerebral hemorrhage using the modified Rankin Scale during follow-up. | 24 months
  Describe the proportion of patients with favorable functional outcome measured with modified Rankin Scale (favorable is the score is 0-2)
Explore vascular mortality and overall mortality in patients with remote cerebral hemorrhage during follow-up. | 24 months
  Describe the frequency, rate and adjusted hazard ratio
Explore cognitive impairment follow-up | 24 months
  IQCODE brief test >56 points

CONTACTS AND LOCATIONS:
Overall Officials: Luis Prats Sanchez, MD PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided